CLINICAL TRIAL: NCT04733261
Title: Effectiveness Of Diaphragmatic Mobility In Ventilated Assisted Patients
Brief Title: Diaphragmatic Mobility In Ventilated Assisted Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical Services (Pvt) Ltd (Industry)
Responsible Party: Principal Investigator, Mir Arif Hussain, Assistant professor, Aqua Medical Services (Pvt) Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rimsha zeb 00568
Record Dates: First submitted 2020-12-22; First posted 2021-02-02 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Ventilation Therapy; Complications
Keywords: Respiration, Artificial; Diaphragm; Physical Therapy Modalities; Ventilators, Mechanical; Intensive Care Units
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic mobility (Active Comparator): The patient will be in supine, supported on one/two pillows under her head, and a bolster under her knees.
  Interventions: Other: Diaphragmatic mobility
- Chest Physiotherapy (Experimental): Give passive ROM exercise to all joints of the upper and lower extremities.
  Interventions: Other: Chest Physiotherapy

INTERVENTIONS:
Other: Diaphragmatic mobility — Therapist will manually make contact with Pisiform Hypothenar region and last three fingers among the underneath the costal cartilage of the 7th in the direction of 10 ribs. For the duration of participant's inhalation, the counselor drag softly within a upward course accompany the increase motion of the ribs. For the period of expiration, the counselor will deepens make contact with in the direction of the internal costal border. Taking place consequent breathing, the counselor wanted on the way to expand traction as well as slickly make deeper the contact.
  Arms: Diaphragmatic mobility
Other: Chest Physiotherapy — Patients allocated to the control group and interventional group received pulmonary rehabilitation two times a day beginning happening the day of entrance on the way to the intensive care unit. It consists of side-lying positioning with the head of the bed horizontal for at least 20 min with the most affected lung on chest x-ray positioned uppermost is also known as postural drainage, 4 sets of 6 cycles of expiratory chest wall vibrations , and airway suctioning at least three times through the endotracheal and tracheotomy tube disperse in the course of the management
  Arms: Chest Physiotherapy

SUMMARY:
The study was a randomized controlled trial. A total of 24 patients who met the inclusion criteria were included in this study and randomly divided by sealed envelope method into Experimental and Control groups with 12 patients each. Assessment of arterial blood gas analyzer (oxygen saturation(SP02), heart rate (HR), respiratory rate(RR), the partial pressure of carbon dioxide(PCO2), the partial pressure of oxygen(PO2), Bicarbonate(HCO3), and potential of hydrogen(PH) and modes of the ventilator (SIMV and PSV) for both groups were carried out at baseline and after 4thsession.The control group was given Chest physiotherapy only. While the Experimental group received Chest physiotherapy with Diaphragmatic Mobility. Total 4 sessions were given on alternate days to both groups.

DETAILED DESCRIPTION:
Most common state in the intensive care unit is an intensive care unit acquired weakness in seriously unwell patients who are artificially ventilated for an extended period of time. The most important aspect of mechanical ventilation in the disuse atrophy and deconditioning of a patient's inspiratory muscle since it can replace the patient's own respiratory muscle exertion. The diaphragm particularly counters to persistent mechanical ventilation with atrophy. Most sufferers who are admitted to an intensive care unit need artificial aeration. Due to weaknesses of respiratory muscle might augment the interval of mechanical ventilation and delay the phase of withdrawal of mechanical ventilation. The term weaning is used for the course of withdrawal of artificial aeration to facilitate the patient's own respiratory muscle effort in the intensive care unit. Ventilation is universal work, linking the entire body, the emotions, the nervous system and organs. The diaphragm is the primary breathing muscle that influencing with its contraction the inspiratory actions. Diaphragmatic breathing is recognized as normal breathing which involves corresponding movement of abdomen, upper and lower ribcage. Furthermore, functionality and sufficient use of the diaphragm muscle requires usual breathing. Thoracic breathing is recognized as unusual breathing that involves aeration from the upper chest, evidence by bigger upper rib cage movement, compare to lower rib cage movement. Weakness possibly will owe an extreme weight on the respiratory muscle, which might affect starting augmented airway conflict and also over-come lung compliance. Two most important factors that are broadly known as a reason of malfunction to with-drawl from mechanical ventilation are weakness or fatigue of diaphragm and accessory muscle of respiration. A dome-shaped muscular membrane that separates the abdomen from thoracic is a diaphragm. Nine hundred centimetre per square area is covert in adults. It is the most important and primary inspiratory muscle and it is able to condense itself to forty per cent as of residual to vital capacity. In fact, a one-sided paralysis of the phrenic nerve generates merely respiratory dysfunction because the stomach has the widespread capacity to functional preserved. The weakness of diaphragm muscle tends to be more worse in patients who are mechanically ventilated for a prolonged period of time with controlled modes of mechanical ventilator compared to spontaneous modes and also appear to be interrelated to patients voluntary inspiratory exertion even as ventilator-dependent. During inspiration, throughout the application of resistance in inspiratory muscles that may help in strengthening of inspiratory muscle and this technique is known as inspiratory muscle training. Patients who have difficulty in breathing and mechanically ventilated for more than 24 hours possibly will adversely affect diaphragmatic structure and function. Major factors such as reduced quality of life, increase the length of stay in the intensive care unit, increase death rate and reduced functional grades are due to extended artificial aeration. Moreover, extended artificial aeration is cheap, unbearable a big portion of hospital assets and a healthcare load that might keep on subsequent hospital ejection. An intervention invented to directly stretch the muscle fibre of diaphragm is known as the manual diaphragm release technique. Even though this intervention is widely used in some regions, there is no quantitative research or systematic trails or evaluating the result of this technique. The previous research conducted to find out the outcome of manual diaphragm release technique in chronic obstructive pulmonary disease. The objective of the study was to determine the effects of diaphragmatic mobility on improving ventilation in ventilated assisted patients, to determine the effects of diaphragmatic mobility in weaning off from mechanical ventilation in ventilated assisted patients, and to determine the additional effects of diaphragmatic mobility on respiration along with Chest Physical Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 60
* Oro-tracheal or nasotracheal intubate; ventilator mode:- Synchronized intermittent mechanical ventilation(SIMV) or Pressure support SIMV
* Both Gender included have been aeration used for Acute Respiratory Failure( type 2) during SIMV/PSV used for at any rate 72 hours consecutively
* Hemodynamically secure with no vasopressin or else inotropes (apart from a dobutamine and dopamine infusion lesser than 5 gamma/Kg/min and a 3 gamma /Kg/min, correspondingly
* Positive end-expiratory pressure 5 to 7cm H2O

Exclusion Criteria:

* Neurological or neuromuscular disorders
* Dysfunction of Phrenic Nerve
* Insertion of a nasogastric tube (for example recent upper gastrointestinal surgery, oesophagal varies).
* Pulmonary embolism, Malignancy, Pneumothorax, trauma, fever
* Acutearrhythmias

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Synchronized Intermittent- Mandatory Ventilation (SIMV) | 0 day
  Synchronized intermittent mandatory ventilation is a ventilator mode that enables partial mechanical assistance. This ventilator mode will provide a set number of breaths at a fixed tidal volume, but a patient can trigger a spontaneous breath with the volume determined by patient effort
Pressure Support Ventilation (PSV) | 0 day
  For the spontaneously breathing patient, pressure support ventilation (PSV) has been advocated to limit barotrauma and to decrease the work of breathing. ... Airway pressure support is maintained until the patient's inspiratory flow falls below a certain cutoff (eg, 25% of peak flow).
Synchronized Intermittent- Mandatory Ventilation (SIMV) | 4th day
  Synchronized intermittent mandatory ventilation is a ventilator mode that enables partial mechanical assistance. This ventilator mode will provide a set number of breaths at a fixed tidal volume, but a patient can trigger a spontaneous breath with the volume determined by patient effort
Pressure Support Ventilation (PSV) | 4th day
  For the spontaneously breathing patient, pressure support ventilation (PSV) has been advocated to limit barotrauma and to decrease the work of breathing. ... Airway pressure support is maintained until the patient's inspiratory flow falls below a certain cutoff (eg, 25% of peak flow).

SECONDARY OUTCOMES:
Arterial Blood Gas ( ABGs) Test | 0 day,4th day
  An arterial-blood gas test measures the amounts of arterial gases, such as oxygen and carbon dioxide. An ABG test requires that a small volume of blood be drawn from the radial artery with a syringe and a thin needle, but sometimes the femoral artery in the groin or another site is used.
Peripheral Capillary Oxygen Saturation (SPO2) | 0 day,4th day
  SpO2 stands for peripheral capillary oxygen saturation, an estimate of the amount of oxygen in the blood. More specifically, it is the percentage of oxygenated haemoglobin (haemoglobin containing oxygen) compared to the total amount of haemoglobin in the blood ( oxygenated and non-oxygenated haemoglobin).
Chest X-ray | 0 day,4th day
  The chest x-ray is the most commonly performed diagnostic x-ray examination. A chest x-ray produces images of the heart, lungs, airways, blood vessels and the bones of the spine and chest.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Abdul Ghafoor Sajjad,, PHD*, Principal Investigator — Shifa Tameer e milat University
Locations (1):
- Aqua research Center, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jounieaux V, Duran A, Levi-Valensi P. Synchronized intermittent mandatory ventilation with and without pressure support ventilation in weaning patients with COPD from mechanical ventilation. Chest. 1994 Apr;105(4):1204-10. doi: 10.1378/chest.105.4.1204. PMID 8162750
- [Background] Hodgson CL, Tipping CJ. Physiotherapy management of intensive care unit-acquired weakness. J Physiother. 2017 Jan;63(1):4-10. doi: 10.1016/j.jphys.2016.10.011. Epub 2016 Nov 26. PMID 27989729
- [Background] Bordoni B, Marelli F, Morabito B, Sacconi B. Manual evaluation of the diaphragm muscle. Int J Chron Obstruct Pulmon Dis. 2016 Aug 18;11:1949-56. doi: 10.2147/COPD.S111634. eCollection 2016. PMID 27574419
- [Background] Moodie L, Reeve J, Elkins M. Inspiratory muscle training increases inspiratory muscle strength in patients weaning from mechanical ventilation: a systematic review. J Physiother. 2011;57(4):213-21. doi: 10.1016/S1836-9553(11)70051-0. PMID 22093119
- [Background] Bissett B, Leditschke IA, Green M, Marzano V, Collins S, Van Haren F. Inspiratory muscle training for intensive care patients: A multidisciplinary practical guide for clinicians. Aust Crit Care. 2019 May;32(3):249-255. doi: 10.1016/j.aucc.2018.06.001. Epub 2018 Jul 11. PMID 30007823
- [Background] Rocha T, Souza H, Brandao DC, Rattes C, Ribeiro L, Campos SL, Aliverti A, de Andrade AD. The Manual Diaphragm Release Technique improves diaphragmatic mobility, inspiratory capacity and exercise capacity in people with chronic obstructive pulmonary disease: a randomised trial. J Physiother. 2015 Oct;61(4):182-9. doi: 10.1016/j.jphys.2015.08.009. Epub 2015 Sep 19. PMID 26386894
- [Background] Nair A, Alaparthi GK, Krishnan S, Rai S, Anand R, Acharya V, Acharya P. Comparison of Diaphragmatic Stretch Technique and Manual Diaphragm Release Technique on Diaphragmatic Excursion in Chronic Obstructive Pulmonary Disease: A Randomized Crossover Trial. Pulm Med. 2019 Jan 3;2019:6364376. doi: 10.1155/2019/6364376. eCollection 2019. PMID 30719351
- [Background] Yang PH, Wang CS, Wang YC, Yang CJ, Hung JY, Hwang JJ, Wang TH, Chuang IC, Huang MS. Outcome of physical therapy intervention on ventilator weaning and functional status. Kaohsiung J Med Sci. 2010 Jul;26(7):366-72. doi: 10.1016/S1607-551X(10)70060-7. PMID 20638039